CLINICAL TRIAL: NCT04818658
Title: The Preformed Metal Crowns Placed Using the Hall Technique Versus the Conventional Restoration: A 5-year Retro-prospective Clinical Study
Brief Title: The Preformed Metal Crowns Placed Using the Hall Technique Versus the Conventional Restoration
Status: Completed | Type: Observational
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Betul Sen Yavuz, Assistant Professor, Bahçeşehir University
Other Study IDs: 441555555
Record Dates: First submitted 2021-03-24; First posted 2021-03-26 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Dental Caries; Caries; Dentin
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Preformed Metal Crowns using Hall Technique
  Interventions: Other: Assessment of the stainless steel crown using the Hall Technique and Compomer Restoration on primary molars
- Compomer Restoration
  Interventions: Other: Assessment of the stainless steel crown using the Hall Technique and Compomer Restoration on primary molars

INTERVENTIONS:
Other: Assessment of the stainless steel crown using the Hall Technique and Compomer Restoration on primary molars — Intra-oral clinical examination is performed and restorations are evaluated by the practitioner. Periapical radiography is taken according to national guidelines.

SUMMARY:
The aim of this study is to compare the survival rate of the conventional restorations with the Hall Technique in carious primary molars.

DETAILED DESCRIPTION:
comparing the survival rate of the conventional restorations with the Hall Technique in carious primary molars.

ELIGIBILITY:
Inclusion Criteria:

* patients aged five to eight years at the time of dental treatment,
* patients attending follow-up appointments
* patients with compomer restoration and Hall restoration in their teeth
* patients with matching the extent of caries in the two groups

Exclusion Criteria:

* patients not attending follow-up appointments
* patients without both treatment

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: patients aged 5-8 years treated with preformed metal crowns using Hall Technique and compomer restoration
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2021-10-03 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
The survival rate of Hall Technique and Compomer Restorations | 5 year
  1. Successful: restoration satisfactory, no additional treatment required, no clinical sign and symptoms of pulpal pathology or tooth exfoliated,
  2. Minor failure: restoration wear/fracture/loss (restorable) or crown perforation, secondary caries or new caries, reversible pulpitis treated without requiring extraction or pulpotomy,
  3. Major failure: the tooth is broken down (unrestorable), inter-radicular radiolucency or internal root resorption, signs or symptoms of irreversible pulpitis requiring extraction or pulpotomy.
  4. The survival analysis: the restorations are assessed as successful or failure.

CONTACTS AND LOCATIONS:
Overall Officials: Betul Sen Yavuz, Principal Investigator — Bahçeşehir University
Locations (1):
- Bahcesehir University, Istanbul, Turkey (Türkiye)